CLINICAL TRIAL: NCT01861444
Title: National, Multicenter, Observational Study Evaluating Prevalence, Virological and Clinical Characteristics of Chronic Hepatitis Delta in Romania and Assess Efficacy of Peg-interferon Alfa-2a Treatment in Patients With Chronic Hepatitis D (CHD)
Brief Title: An Observational Study on the Prevalence of Chronic Hepatitis D in Romania and the Efficacy of Treatment With Pegasys (Peginterferon Alfa-2a)
Status: Terminated | Type: Observational
Why Stopped: Terminated due to financial reasons.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25581
Record Dates: First submitted 2013-05-02; First posted 2013-05-23 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis D, Chronic
MeSH Terms: conditions — Hepatitis D, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective, multicenter, observational study will assess the prevalence of chronic hepatitis D in patients with chronic hepatitis B in Romania and evaluate the efficacy of Pegasys (peginterferon alfa-2a) in patients with chronic hepatitis D. Eligible patients treated with Pegasys according to current medical practice will be followed until 24 weeks after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

For epidemiological part of the study:

* Adult patients >/= 18 years of age
* Positive HBsAg for at least 6 months

For the non-interventional section of the study

* Adult patients, >/= 18 years of age
* Positive HBsAg for at least 6 months
* Positive anti-delta and positive HDV RNA by PCR
* Elevated serum ALT >/= 2x ULN

Exclusion Criteria:

Patients with any of the following will not be eligible for treatment with Pegasys:

* History of neurological disease
* History of severe psychiatric disease
* Decompensated diabetes
* History of immunologically mediated disease
* History of severe cardiac disease
* History or other evidence of severe chronic pulmonary disease
* Inadequate hematologic function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis B, and then those who are positive for anti-HDV Ab and treated with Pegasys
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2011-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Proportion of chronic hepatitis B patients in Romania with chronic hepatitis D infection | approximately 3.5 years
Response rate: Proportion of patients achieving ALT normalization and HDV RNA negativity 24 weeks after the end of treatment | approximately 3.5 years

SECONDARY OUTCOMES:
Virological characteristics (HBeAg/anti-HBe/HBV DNA/anti-HDV Ab/HDV RNA) of patients with chronic hepatitis D | approximately 3.5 years
Proportion of chronic hepatitis D patients with liver cirrhosis | approximately 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Bucharest, Romania